CLINICAL TRIAL: NCT00827112
Title: Pilot Study Of Novel Combination Of Maraviroc + Atazanavir/Ritonavir vs. Atazanavir/Ritonavir + Emtricitabine/Tenofovir For The Treatment Of Naïve HIV-Infected Patients With R5 HIV-1
Brief Title: A Pilot Study Of A Novel Treatment Regimen, Maraviroc + Ritonavir Boosted Atazanavir, In Treatment Naive HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4001078
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Human Immunodeficiency Virus-1
Keywords: CCR5-tropic HIV-1 virus
MeSH Terms: interventions — Maraviroc; Lopinavir; lopinavir-ritonavir drug combination; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): maraviroc (Selzentry, Celsentri) 150 mg QD + atazanavir (Reyataz) /ritonavir (Norvir) 300/100mg QD Subjects experiencing unconjugated hyperbilirubinemia attributable to atazanavir (Reyataz) /ritonavir (Norvir) without any other etiology of hyperbilirubinemia, responding to the therapy without virologic failure, but expressing cosmetic concerns because of the jaundice or scleral icterus (associated with bilirubin elevations) and wish to discontinue atazanavir (Reyataz) in spite of reassurances by the investigator, will be permitted on a single occasion only to switch to another protease inhibitor either darunavir (Prezista)/ritonavir (Norvir)((800/100 mg) QD or lopinavir/ritonavir (Kaletra, Aluvia)(400/100mg) BID and remain in the study. If the investigator decides to switch to a protease inhibitor other than darunavir (Prezista)/ritonavir (Norvir) or lopinavir/ritonavir (Kaletra, Aluvia)(, then the subject must be discontinued from the study.
  Interventions: Drug: maraviroc
- Arm B (Experimental): emtricitabine/tenofovir (Truvada) 200/300mg QD + atazanavir (Reyataz) /ritonavir (Norvir) 300/100 mg QD
  Subjects experiencing unconjugated hyperbilirubinemia attributable to atazanavir (Reyataz) /ritonavir (Norvir) without any other etiology of hyperbilirubinemia, responding to the therapy without virologic failure, but expressing cosmetic concerns because of the jaundice or scleral icterus (associated with bilirubin elevations) and wish to discontinue atazanavir in spite of reassurances by the investigator, will be permitted on a single occasion only to switch to another protease inhibitor either darunavir/ritonavir (800/100 mg) QD or lopinavir/ritonavir (400/100mg) BID and remain in the study. If the investigator decides to switch to a protease inhibitor other than darunavir/ritonavir or lopinavir/ritonavir, then the subject must be discontinued from the study.
  Interventions: Drug: maraviroc

INTERVENTIONS:
Drug: maraviroc — maraviroc (Selzentry, Celsentri) 150mg QD + atazanavir (Reyataz) /ritonavir (Norvir) (300/100mg) QD OR maraviroc (Selzentry, Celsentri) 150mg QD+ darunavir (Prezista)/ritonavir (Norvir) (800/100 mg) QD (if atazanavir (Reyataz) /ritonavir (Norvir) is replaced by darunavir (Prezista)/ritonavir (Norvir)) OR maraviroc (Selzentry, Celsentri) 150mg QD+ lopinavir/ritonavir (Kaletra, Aluvia) (400/100 mg) BID (if atazanavir (Reyataz) /ritonavir (Norvir) is replaced by lopinavir/ritonavir (Kaletra, Aluvia))
  Other Names: maraviroc =Celsentri, Selzentry; atazanavir =Reyataz; ritonavir =Norvir; lopinavir/ritonavir=Kaletra, Aluvia; darunavir=Prezista
  Arms: Arm A
Drug: maraviroc — emtricitabine/tenofovir (Truvada) 200/300mg QD + atazanavir (Reyataz) /ritonavir (Norvir) 300/100 mg QD OR emtricitabine/tenofovir (Truvada) 200/300 mg QD + darunavir (Prezista)/ritonavir (Norvir) (800/100 mg) QD (if atazanavir (Reyataz) /ritonavir (Norvir) is replaced by darunavir (Prezista)/ritonavir (Norvir)) OR emtricitabine/tenofovir (Truvada) 200/300 mg QD + lopinavir/ritonavir(Kaletra, Aluvia) (400/100 mg) BID (if atazanavir (Reyataz) /ritonavir (Norvir) is replaced by lopinavir/ritonavir (Kaletra, Aluvia))
  Other Names: maraviroc=Celsentri, Selzentry; emtricitabine/tenofovir=Truvada; atazanavir =Reyataz; ritonavir =Norvir; lopinavir/ritonavir=Kaletra, Aluvia
  Arms: Arm B

SUMMARY:
This is a pilot study to examine if the novel treatment regimen maraviroc plus boosted atazanavir can be expected to be safe and efficacious in treatment naive HIV infected patients. Based on the results from this study, a confirmatory phase 3 study may be conducted.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA viral load of ≥1,000 copies/mL measured at the Screening Visit.
* CD4 count ≥100 cells/mm3 at Screening.
* Have only R5 HIV-1 at Screening as verified by the Monogram Bioscience Trofile® assay with enhanced sensitivity.

Exclusion Criteria:

* Prior treatment with any other HIV antiretroviral therapy for more than 14 days at any time.
* Any evidence of resistance to atazanavir, tenofovir, and emtricitabine.
* X4-or dual/mixed-tropic virus by enhanced Trofile assay or repeated assay failure or not reportable results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (19):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Addison, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Spokane, Washington
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, München
- Spain (6):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001078&StudyName=A%20Pilot%20Study%20Of%20A%20Novel%20Treatment%20Regimen%2C%20Maraviroc%20+%20Ritonavir%20Boosted%20Atazanavir%2C%20In%20Treatment%20Naive%20HIV-Infected%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc+ Atazanavir / Ritonavir: Maraviroc 150 milligram (mg) tablets once daily along with atazanavir/ritonavir 300 mg/100 mg tablets once daily were orally administered for 96 weeks.
- Atazanavir / Ritonavir + Emtricitabine / Tenofovir: Atazanavir/ritonavir 300 mg/100 mg tablets once daily along with emtricitabine/tenofovir 200 mg/245 mg tablets once daily were orally administered for 96 weeks.
Period: Overall Study
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Started | 65 | 64
Treated | 60 | 61
Completed | 50 | 52
Not Completed | 15 | 12
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Randomized but not treated | 5 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir | Total
Number analyzed (Participants) | 60 | 61 | 121
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (10.2) | 35.3 (10.5) | 36.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 56 | 52 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immuno Deficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) Levels Less Than 50 Copies/Milliliter (mL)
Time Frame: Week 48
Population: Full Analysis Set (FAS) population included those participants who had taken at least one dose of the study drug, had baseline and at least one post baseline measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Percentage of participants | 74.60 [63.47 to 85.69] | 83.60 [74.32 to 92.90]

2. Secondary Outcome: HIV-1 RNA Levels at Baseline
Time Frame: Baseline
Population: FAS population included those participants who had taken at least one dose of the study drug, had baseline and at least one post baseline measurement.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
copies/mL | 84982 (127008) | 114827 (149638)

3. Secondary Outcome: Change From Baseline in HIV-1 RNA Levels of First 15 Participants at Days 4, 7, 10 and 14
Description: Plasma HIV-1 RNA levels were evaluated for first 15 participants enrolled at United States (U.S) sites only.
Time Frame: Baseline , Days 4, 7, 10 and 14
Population: First 15 participants who were enrolled at U.S sites and had taken the study drug .
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 14 | 16
copies/mL
  Change at Day 4 | 1800.00 (37351.09) | -46479.40 (62259.15)
  Change at Day 7 | -36947.90 (28463.80) | -52137.10 (68684.14)
  Change at Day 10 | -58595.80 (66157.66) | -54925.90 (70846.93)
  Change at Day 14 | -47271.60 (38234.34) | -55449.90 (71207.16)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Maraviroc
Time Frame: Day 14 (0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose)
Population: Pharmacokinetic (PK) parameter analysis population included first 15 participants treated with maraviroc.
Measure: Median (Full Range); unit: nanogram (ng)/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir
Number analyzed (Participants) | 15
nanogram (ng)/mL | 650 [178 to 1490]

5. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Maraviroc
Time Frame: Day 14 (0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose)
Population: PK parameter analysis population included first 15 participants treated with maraviroc.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir
Number analyzed (Participants) | 15
ng/mL | 37.0 [8.4 to 92.7]

6. Secondary Outcome: Average Observed Plasma Concentration (Cavg) of Maraviroc
Description: Cavg was described as area under the plasma concentration-time profile from time zero to time 24 hours (AUC24) divided by the dosing interval (AUC24/ 24).
Time Frame: Day 14 (0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose)
Population: PK parameter analysis population included first 15 participants treated with maraviroc.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir
Number analyzed (Participants) | 15
ng/mL | 185.10 (71.08)

7. Secondary Outcome: Change From Baseline in Plasma log10 Viral Load at Weeks 16, 24, 48 and 96
Time Frame: Baseline, Week 16, Week 24, Week 48, Week 96
Population: FAS population included those participants who had taken at least one dose of the study drug, had a baseline and at least one post baseline measurement. Here "n" signified participants who received the study drug and evaluated at the time point.
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
log10 copies/ml
  Baseline (n= 59, 61) | 84982 (127008) | 114827 (149638)
  Change at Week 16 (n= 54, 58) | -89859.1 (131317.35) | -107684.6 (149476.47)
  Change at Week 24 (n= 56, 58) | -87241.2 (129638.57) | -110498.1 (149836.29)
  Change at Week 48 (n= 53, 54) | -82343.4 (119356.62) | -115582.9 (153705.26)
  Change at Week 96 (n= 49, 51) | -80117.7 (121443.50) | -99662.6 (116525.87)

8. Secondary Outcome: Percentage of Participants With Less Than 50 Copies/mL of HIV-1 RNA
Time Frame: Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Percentage of participants
  Week 2 (n= 55, 60) | 0 [0 to 0] | 6.60 [0.35 to 12.77]
  Week 4 (n= 57, 60) | 8.50 [1.37 to 15.58] | 21.30 [11.03 to 31.59]
  Week 8 (n= 57, 59) | 47.50 [34.72 to 60.20] | 42.60 [30.21 to 55.03]
  Week 12 (n= 55, 59) | 61.00 [48.57 to 73.46] | 62.30 [50.13 to 74.46]
  Week 16 (n= 54, 58) | 72.90 [61.54 to 84.23] | 73.80 [62.73 to 84.81]
  Week 20 (n= 56, 57) | 71.20 [59.63 to 82.74] | 83.61 [74.32 to 92.90]
  Week 24 (n= 56, 58) | 81.36 [71.42 to 91.29] | 88.52 [80.53 to 96.52]
  Week 32 (n= 55, 57) | 79.66 [69.39 to 89.93] | 88.52 [80.53 to 96.52]
  Week 40 (n= 54, 55) | 81.36 [71.42 to 91.29] | 88.52 [80.53 to 96.52]
  Week 48 (n= 53, 54) | 74.58 [63.47 to 85.69] | 83.61 [74.32 to 92.90]
  Week 60 (n= 52, 53) | 67.80 [55.87 to 79.72] | 85.25 [76.35 to 94.15]
  Week 72 (n= 52, 53) | 74.58 [63.47 to 85.69] | 81.97 [72.32 to 91.62]
  Week 84 (n= 50, 52) | 76.27 [65.42 to 87.13] | 83.61 [74.32 to 92.90]
  Week 96 (n= 49, 51) | 67.80 [55.87 to 79.72] | 81.97 [72.32 to 91.62]

9. Secondary Outcome: Percentage of Participants With Less Than 400 Copies/mL of HIV-1 RNA
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Percentage of participants
  Week 2 (n= 55, 60) | 27.12 [15.77 to 38.46] | 34.43 [22.50 to 46.35]
  Week 4 (n= 57, 60) | 50.85 [38.09 to 63.60] | 52.46 [39.93 to 64.99]
  Week 8 (n= 57, 59) | 79.66 [69.39 to 89.93] | 77.05 [66.50 to 87.60]
  Week 12 (n= 55, 59) | 89.83 [82.12 to 97.54] | 88.52 [80.53 to 96.52]
  Week 16 (n= 54, 58) | 88.14 [79.88 to 96.39] | 91.80 [84.92 to 98.69]
  Week 20 (n= 56, 57) | 89.83 [82.12 to 97.54] | 93.44 [87.23 to 99.65]
  Week 24 (n= 56, 58) | 91.53 [84.42 to 98.63] | 93.44 [87.23 to 99.65]
  Week 32 (n= 55, 57) | 89.83 [82.12 to 97.54] | 93.44 [87.23 to 99.65]
  Week 40 (n= 54, 55) | 91.53 [84.42 to 98.63] | 90.16 [82.69 to 97.64]
  Week 48 (n= 53, 54) | 89.83 [82.12 to 97.54] | 86.89 [78.41 to 95.36]
  Week 60 (n= 52, 53) | 86.44 [77.70 to 95.18] | 86.89 [78.41 to 95.36]
  Week 72 (n= 52, 53) | 86.44 [77.70 to 95.18] | 85.25 [76.35 to 94.15]
  Week 84 (n= 50, 52) | 81.36 [71.42 to 91.29] | 85.25 [76.35 to 94.15]
  Week 96 (n= 49, 51) | 77.97 [67.39 to 88.54] | 83.61 [74.32 to 92.90]

10. Secondary Outcome: Time to Loss of Virological Response (TLOVR)
Description: TLOVR (virological failure) was defined as the time from first dose of study treatment (Day 1) until the time of virologic failure using the time to loss of virologic response algorithm.
Time Frame: Baseline through Week 96
Population: FAS population included those participants who had taken at least one dose of the study drug, had a baseline and at least one post baseline measurement.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Days | 436.2 (22.5) | 463.8 (16.1)

11. Secondary Outcome: Time-Averaged Difference (TAD) in log10 Viral Load
Description: TAD was calculated as area under the curve of HIV divided by time period minus baseline HIV where HIV was denoted as HIV-1 RNA (log10 copies/mL).
Time Frame: Week 16, Week 24, Week 48, Week 96
Population: FAS population included those participants who had taken at least one dose of the study drug, had a baseline and at least one post baseline measurement. Here N (Number of participants analyzed) signified participants evaluable for the measure.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 51 | 52
log10 copies/mL
  Week 16 | -2.459 (0.046) | -2.402 (0.045)
  Week 24 | -2.663 (0.048) | -2.626 (0.046)
  Week 48 | -2.897 (0.046) | -2.868 (0.050)
  Week 96 | -2.998 (0.055) | -3.001 (0.053)

12. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+T Lymphocyte (CD4) Cell Counts at Weeks 16, 24, 48 and 96
Time Frame: Baseline, Week 16, Week 24, Week 48, Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/microliter (cells/mcL)
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
cells/microliter (cells/mcL)
  Baseline (n= 59, 61) | 357.70 (123.53) | 390.00 (152.34)
  Change at Week 16 (n= 54, 58) | 169.60 (117.20) | 139.80 (102.62)
  Change at Week 24 (n= 54, 57) | 188.90 (125.14) | 173.30 (130.55)
  Change at Week 48 (n= 52, 53) | 215.70 (166.59) | 226.60 (138.04)
  Change at Week 96 (n= 50, 51) | 287.50 (173.23) | 298.50 (160.54)

13. Secondary Outcome: Change From Baseline in Cluster of Differentiation 8+T Lymphocyte (CD8) Cell Count at Weeks 16, 24, 48 and 96
Time Frame: Baseline, Week 16, Week 24, Week 48, Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
cells/mcL
  Baseline (n= 59, 61) | 931.10 (446.26) | 1125.60 (735.08)
  Change at Week 16 (n= 54, 58) | 63.70 (290.49) | -153.80 (473.96)
  Change at Week 24 (n= 54, 57) | 6.20 (334.89) | -178.00 (508.75)
  Change at Week 48 (n= 52, 53) | -76.80 (354.48) | -267.60 (574.22)
  Change at Week 96 (n= 50, 51) | -63.00 (355.60) | -231.40 (516.99)

14. Secondary Outcome: Number of Participants With Genotypic Resistance
Description: Genotypic resistance was assessed for all participants at screening and was evaluated for protease inhibitors (PIs), Nucleotide reverse transcriptase inhibitors (NRTIs), and non-NRTIs (NNRTIs) using Monogram GenoSeq and/or PhenoSenseGT assays. This was then repeated for all participants with HIV-1 viral load more than 500 copies/mL either at treatment failure or at early termination, up to Week 96.
Time Frame: Week 96 or Time of treatment failure
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Phenotypic Resistance
Description: Phenotypic resistance was assessed for all participants at screening and was evaluated for PIs, NRTIs, and NNRTIs using Monogram GenoSeq and/or PhenoSenseGT assays. This was then repeated for all participants with HIV-1 viral load more than 500 copies/mL either at treatment failure or at early termination, up to Week 96.
Time Frame: Week 96 or Time of treatment failure
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 59 | 61
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With HIV-1 RNA Tropism Status Using Trofile Assay
Description: Viral tropism was determined using the trofile assay with enhanced sensitivity for participants with HIV-1 RNA greater than equal to 1000 copies/mL. The enhanced trofile assay had the sensitivity to detect 100 percent of spiked samples when C-X-C chemokine receptor type 4 {CXCR4} [X4]-using HIV-1 RNA represented 0.3 percent of the total viral population.
Time Frame: Baseline to Week 96 or Time of treatment Failure
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine / Tenofovir
Number analyzed (Participants) | 60 | 61
Participants
  Baseline | 60 | 61
  Week 96 or Time of treatment Failure | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to follow-up period (28 days after the last dose of study)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Maraviroc+ Atazanavir / Ritonavir: Maraviroc 150 milligram (mg) tablets once daily along with atazanavir 300 mg or ritonavir 100 mg tablets once daily were orally administered for 96 weeks.
- Atazanavir / Ritonavir + Emtricitabine/ Tenofovir: Atazanavir/ritonavir 300 mg/100 mg tablets QD along with emtricitabine/tenofovir 200 mg/245 mg tablets once daily were orally administered for 96 weeks.
Arm/Group | Maraviroc+ Atazanavir / Ritonavir | Atazanavir / Ritonavir + Emtricitabine/ Tenofovir
Serious Adverse Events (participants affected / at risk) | 13/60 | 11/61
Other Adverse Events (participants affected / at risk) | 55/60 | 58/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc+ Atazanavir / Ritonavir (N=60) | Atazanavir / Ritonavir + Emtricitabine/ Tenofovir (N=61)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anogenital warts (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Parotitis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc+ Atazanavir / Ritonavir (N=60) | Atazanavir / Ritonavir + Emtricitabine/ Tenofovir (N=61)
Ocular icterus (Eye disorders) | 13 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 14
Haemorrhoids (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 6 | 16
Vomiting (Gastrointestinal disorders) | 8 | 6
Fatigue (General disorders) | 3 | 7
Pyrexia (General disorders) | 4 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 18 | 16
Jaundice (Hepatobiliary disorders) | 10 | 6
Anogenital warts (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 8 | 5
Gonorrhoea (Infections and infestations) | 4 | 2
Herpes zoster (Infections and infestations) | 3 | 6
Influenza (Infections and infestations) | 4 | 6
Nasopharyngitis (Infections and infestations) | 3 | 6
Sinusitis (Infections and infestations) | 10 | 3
Tonsillitis (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8
Aspartate aminotransferase increased (Investigations) | 4 | 1
Blood amylase increased (Investigations) | 4 | 2
Blood bilirubin increased (Investigations) | 7 | 5
Blood creatine phosphokinase increased (Investigations) | 6 | 0
Blood creatinine increased (Investigations) | 3 | 1
Blood uric acid increased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 9
Depression (Psychiatric disorders) | 7 | 8
Insomnia (Psychiatric disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Conjunctivitis (Eye disorders) | 1 | 5
Pharyngitis (Infections and infestations) | 3 | 3
Syphilis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Alanine aminotransferase increased (Investigations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.